CLINICAL TRIAL: NCT02799862
Title: A Non-interventional Study of Nab-paclitaxel (Abraxane®) in Combination With Carboplatin as First Line Therapy in Patients With Advanced Non-small Cell Lung Cancer (NEPTUN)
Brief Title: Nab-Paclitaxel in Combination With Carboplatin as First-line Therapy in Patients With NSCLC
Acronym: NEPTUN
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-110333
Record Dates: First submitted 2016-04-29; First posted 2016-06-15 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: metastatic; locally advanced; unresectable; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered in accordance with the SmPC of Nab-Paclitaxel.
  Other Names: Abraxane
Drug: Carboplatin — Carboplatin will be administered as combination partner of Nab-Paclitaxel in accordance with SmPC of Nab-Paclitaxel.

SUMMARY:
This is a single-arm non-interventional study (NIS) to evaluate the effectiveness, safety and quality of life (QoL) in patients with advanced NSCLC receiving the combination of nab-paclitaxel and carboplatin as first line palliative therapy in a real life setting.

DETAILED DESCRIPTION:
The present NIS is designed to provide additional knowledge in terms of effectiveness, safety and quality of life in routine administration of the combination of nab-paclitaxel (Abraxane®) and carboplatin as first line treatment for adult patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who are not candidates for potentially curative surgery and / or radiation therapy. The combination of Abraxane® and carboplatin has been approved in Europe in March 2015 based on results from a pivotal randomized, open label phase III study with 1,052 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of locally advanced / metastatic, unresectable NSCLC
* According to SmPC

Exclusion Criteria:

* According to SmPC

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with locally advanced / metastatic NSCLC who are not candidates for potentially curative surgery and / or radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate | After 6-months
  Effectiveness in terms of PFS will be assessed and evaluated according to local medical standards from screening until end of treatment observation (6 months). Additional survival and and if applicable clinical PFS will be followed up for 24 months post-treatment observation.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | After 6-months
  Effectiveness in terms of OS will be assessed and evaluated according to local medical standards from screening until end of treatment observation (6 months).
Overall Response Rate (ORR) | After 6-months
  Effectiveness in terms of ORR will be assessed and evaluated according to local medical standards from screening until end of treatment observation (6 months).
Safety - Adverse events (AEs) | through study completion, an average of 9 months
  Safety assessments will consist of monitoring of all AEs, including serious adverse events, and monitoring of laboratory values. AEs will be graded according to CTCAE V4.03. Supportive therapies will be documented.
Patient-reported outcomes on Quality of Life | Baseline, after 6 weeks, after 3 months, every 3 months throughout study completion, an average of 9 months
  Questionnaires: EQ5D-5L and FACT-L
Rationale for physicians' treatment decision | Baseline
  Rationale for physicians' treatment decision, assessed with a therapy-decision questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dechow, Prof. Dr., Principal Investigator — Oncology Ravensburg
Locations (1):
- iOMEDICO, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Warmerdam LJ, Rodenhuis S, ten Bokkel Huinink WW, Maes RA, Beijnen JH. The use of the Calvert formula to determine the optimal carboplatin dosage. J Cancer Res Clin Oncol. 1995;121(8):478-86. doi: 10.1007/BF01218365. PMID 7642691
- [Background] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Reck M, Popat S, Reinmuth N, De Ruysscher D, Kerr KM, Peters S; ESMO Guidelines Working Group. Metastatic non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii27-39. doi: 10.1093/annonc/mdu199. Epub 2014 Aug 11. No abstract available. PMID 25115305
- [Background] Gelderblom H, Verweij J, Nooter K, Sparreboom A. Cremophor EL: the drawbacks and advantages of vehicle selection for drug formulation. Eur J Cancer. 2001 Sep;37(13):1590-8. doi: 10.1016/s0959-8049(01)00171-x. PMID 11527683
- [Derived] Dechow T, Riera-Knorrenschild J, Hackanson B, Janssen J, Schulz H, Oppermann U, Chiabudini M, von Weikersthal LF, Budweiser S, Nacke A, Taeuscher D, Welslau M, Potthoff K. First-line nab-paclitaxel plus carboplatin for patients with advanced non-small cell lung cancer: Final results of the NEPTUN study. Int J Cancer. 2023 Jul 1;153(1):141-152. doi: 10.1002/ijc.34467. Epub 2023 Mar 8. PMID 36757197